CLINICAL TRIAL: NCT04075994
Title: A Mobile Relational Agent to Enhance Atrial Fibrillation Self-care
Brief Title: Atrial Fibrillation Health Literacy and Information Technology Trial
Acronym: AFibLITT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Northeastern University (Other); Boston University (Other)
Responsible Party: Principal Investigator, Jared W Magnani, MD, MSc, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY18110147; R61HL144669 (NIH)
Record Dates: First submitted 2019-08-28; First posted 2019-09-03 (Actual); Results first posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Familial Atrial Fibrillation; Arrythmia, Cardiac; Heart Diseases; Pathologic Processes
Keywords: Quality of Life (QoL); Adherence; Health Literacy
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Heart Diseases; Pathologic Processes | interventions — Heart Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Receive the relational agent coupled with the AliveCor Kardia heart rate and rhythm monitor for 120-day use.
  Interventions: Behavioral: Relational Agent and heart rate and rhythm monitor
- Usual care arm (Active Comparator): Receive a brochure on atrial fibrillation, the WebMD app and the AliveCor Kardia heart rate and rhythm monitor for 120-day use.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Relational Agent and heart rate and rhythm monitor — Use of the Relational Agent and heart rate and rhythm monitor daily for 120 days.
  Arms: Intervention arm
Behavioral: Usual Care — Use of the WebMD app and heart rate and rhythm monitor daily for 120 days.
  Arms: Usual care arm

SUMMARY:
Atrial fibrillation (AF) is a common, morbid condition with increasing prevalence. Poor health-related quality of life is common in AF. Patients experience debilitating symptoms and challenging adherence to long-term (possibly lifelong) anticoagulation. The increased risks of stroke, heart failure and mortality associated with AF persist even with optimal treatment. Morbidity in AF is further exacerbated by social factors. Limited health literacy carries challenges of learning a specialized terminology and navigating specialized treatments. In multiple cardiovascular diseases, self-care has demonstrated improvement in self-efficacy, health-related quality of life, symptom burden, and health care utilization - essential components of patient success with AF. Selfcare can provide the critical skills to navigate a challenging chronic disease and improve patient-centered outcomes. Delivery of self-care as a mobile health intervention can complement standard care with a longitudinal intervention to improve patient-centered strategies for AF. While self-care interventions for AF have focused foremost on self-monitoring of anticoagulation,self-care has demonstrated its potential to meet the "triple aim" of improved patient experience, reduced health care utilization, and lower costs.

DETAILED DESCRIPTION:
This is a randomized clinical trial to evaluate the effect of a smartphone-based intervention called a relational agent on health outcomes in people with atrial fibrillation. The study will enroll 240 patients who reside in Pittsburgh-area with this condition and will randomize them to the intervention or control. Intervention participants will receive a smartphone with the agent, which simulates conversation. In addition they will receive an AliveCor Kardia for heart rate and rhythm monitoring, an FDA-approved, widely used instrument that pairs with the smartphone. Control participants will receive a smartphone with WebMD, a brochure published by the American Heart Association that describes AF, and an AliveCor Kardia. The intervention will last 4 months and participants will have visits at baseline, 4, 8 and 12 months. The study will evaluate the improvement in quality of life, medical adherence and health care utilization resulting from the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, age ≥21;
2. Diagnosis of AF, identified from the electronic health record problem list and confirmed by 2 or more reports of AF from separate monitoring events at least 2 weeks apart (electrocardiogram, Holter or event monitor);
3. CHA2DS2-VASc (heart failure, hypertension, age, diabetes, prior stroke or transient ischemic attack, coronary heart disease, female sex)≥2;
4. Prescribed use of warfarin or direct-acting oral anticoagulant for AF stroke prevention;
5. English-speaking well enough to participate in informed consent and this study;
6. No plans to relocate from the area within 12 months of enrollment.

Exclusion Criteria:

1. Conditions other than AF that require anticoagulation, such as mechanical prosthetic valve, deep vein thrombosis, or pulmonary embolism;
2. History of pulmonary vein isolation or foreseen pulmonary vein isolation;
3. History of atrioventricular nodal ablation or foreseen atrioventricular nodal ablation;
4. Heart failure necessitating hospital admission ≤3 months prior to study inclusion;
5. Acute coronary syndrome (defined as at least 2 of the following: chest pain, ischemic electrocardiographic changes, or troponin ≥0.1 ng/mL) ≤3 months prior to study inclusion;
6. Untreated hyperthyroidism or ≤3 months euthyroidism before inclusion;
7. Foreseen pacemaker, internal cardioverter defibrillator, or cardiac resynchronization therapy;
8. Cardiac surgery ≤3 months before inclusion;
9. Planned cardiac surgery;
10. Presence of non-cardiovascular conditions likely to be fatal within 12 months (e.g., cancer);
11. Inability to comprehend the study protocol, defined as failing to answer correctly a set of questions on orientation and short-term memory during the consent process.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jared W Magnani, MD, MSc, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The study team will share individual participant data that underlie the results reported in the study's central manuscripts after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Such data will be available beginning 9 months and ending 36 months following publication of the main manuscripts resulting from this clinical trial.
Access Criteria: Data will be made available to those investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. Proposals may be submitted up to 36 months following article publication. Applicants requesting access to the data will be responsible for the minimal administrative costs to provide the data set.

REFERENCES:
- [Derived] Magnani JW, Lalama CM, Abebe KZ, Ferry D, Rollman BL, Lancet MQ, Kimani E, Olafsson S, Bickmore T, Paasche-Orlow MK. A mobile relational agent to enhance atrial fibrillation self-care: Primary and secondary outcomes of a randomized controlled trial. Am Heart J. 2025 Dec;290:115-128. doi: 10.1016/j.ahj.2025.06.009. Epub 2025 Jun 20. PMID 40545207
- [Derived] Althouse AD, Abebe KZ, Paasche-Orlow MK, Lalama CM, Ferry D, Lancet M, Swabe G, Bickmore T, Magnani JW. Design, rationale, and baseline characteristics of a randomized controlled trial evaluating a mobile relational agent to enhance atrial fibrillation self-care. Contemp Clin Trials. 2023 Jan;124:107015. doi: 10.1016/j.cct.2022.107015. Epub 2022 Nov 17. PMID 36402276

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Receive the relational agent coupled with the AliveCor Kardia heart rate and rhythm monitor for 120-day use.
  Relational Agent and heart rate and rhythm monitor: Use of the Relational Agent and heart rate and rhythm monitor daily for 120 days.
- Usual Care: Receive a brochure on atrial fibrillation, the WebMD app and the AliveCor Kardia heart rate and rhythm monitor for 120-day use.
  Usual Care: Use of the WebMD app and heart rate and rhythm monitor daily for 120 days.
Period: Overall Study
Arm/Group | Intervention | Usual Care
Started | 123 | 120
Completed | 110 | 108
Not Completed | 13 | 12
Not completed — Withdrawal by Subject | 8 | 9
Not completed — Adverse Event | 2 | 2
Not completed — Investigator withdrew | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 123 | 120 | 243
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 71.9 [67.0 to 77.9] | 71.3 [64.1 to 77.0] | 71.7 [66.1 to 77.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 69 | 156
  Male | 36 | 51 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 123 | 117 | 240
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 36 | 38 | 74
  White | 84 | 77 | 161
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 2 | 2
Marital Status [Count of Participants; unit: Participants]
  Never married/never lived as married | 21 | 23 | 44
  Married or living as such | 62 | 59 | 121
  Separated or divorced | 15 | 18 | 33
  Widowed | 25 | 20 | 45
Employment Status [Count of Participants; unit: Participants]
  Working now, full time | 13 | 14 | 27
  Working now, part time | 7 | 5 | 12
  Employed but temporarily laid off | 1 | 1 | 2
  Sick or on leave for health reasons | 3 | 3 | 6
  Unemployed, looking for work | 0 | 1 | 1
  Unemployed, not looking for work | 3 | 8 | 11
  Homemaker, not working outside the home | 3 | 2 | 5
  Retired from my usual job and not working | 82 | 77 | 159
  Retired from my usual job but working for pay | 11 | 9 | 20
Total family income [Count of Participants; unit: Participants]
  Less than or equal to $19,999 | 17 | 12 | 29
  $20,000 to $34,999 | 15 | 20 | 35
  $35,000 to $49,999 | 14 | 18 | 32
  $50,000 to $74,999 | 22 | 17 | 39
  $75,000 to $99,999 | 14 | 13 | 27
  Greater than or equal to $100,000 | 16 | 18 | 34
  Don't know | 13 | 9 | 22
  Prefer not to respond | 12 | 13 | 25
Education [Count of Participants; unit: Participants]
  Some high school with no certificate | 3 | 4 | 7
  High school graduate | 22 | 25 | 47
  Some vocational/trade school with no certificate | 3 | 2 | 5
  Vocational/trade certificate | 6 | 7 | 13
  Some college with no degree | 20 | 22 | 42
  Associate degree | 15 | 15 | 30
  Bachelor degree | 20 | 17 | 37
  Graduate/professional school | 29 | 21 | 50
  Unknown | 5 | 7 | 12
Type of medical insurance [Count of Participants; unit: Participants]
  None | 0 | 1 | 1
  Medicaid | 3 | 1 | 4
  Medicare | 13 | 12 | 25
  Private | 32 | 36 | 68
  Other | 0 | 1 | 1
  Medicaid/Medicare | 11 | 8 | 19
  Medicaid/Tricare | 1 | 0 | 1
  Medicaid/Private | 2 | 1 | 3
  Medicare/Tricare | 0 | 1 | 1
  Medicare/Private | 52 | 55 | 107
  Medicare/Other | 1 | 2 | 3
  Tricare/Private | 1 | 0 | 1
  Private/Other | 1 | 0 | 1
  Great than 2 types | 6 | 2 | 8
Approximate years with Atrial Fibrillation [Median (Inter-Quartile Range); unit: years] | 4 [2 to 10] | 4 [1.5 to 10] | 4 [2 to 10]
Warfarin or Direct-acting oral anticoagulant [Count of Participants; unit: Participants]
  Warfarin (also called Coumadin, Jantoven) | 19 | 15 | 34
  Xarelto (Rivaroxaban) | 30 | 23 | 53
  Pradaxa (Dabigatran) | 1 | 1 | 2
  Eliquis (Apixaban) | 73 | 81 | 154
Non-adherence to oral anticoagulation [Count of Participants; unit: Participants] — Self-reported daily adherence to oral anticoagulation dichotomized as adherent or non-adherent. Three-item instrument each scaled 1-5. Individuals reporting 1 for all items classified as adherent; any individual reporting 2 or higher on any item classified as non-adherent.
  Participants
    Yes | 16 | 17 | 33
    No | 107 | 103 | 210
AF Effect on Quality of Life [Median (Inter-Quartile Range); unit: units on a scale] — AF Effect on Quality-of-Life questionnaire (AFEQT)
  Overall score and individual domain scores at baseline. Scores for the overall score and each subscale range from 0-100. For the overall score and the domains, a score of 0 corresponds to complete disability (or responding "extremely" limited, difficult or bothersome to all questions answered), while a score of 100 corresponds to no disability (or responding "not at all" limited, difficult or bothersome to all questions answered).
  units on a scale
    Overall Score | 74.1 [60.2 to 89.8] | 73.6 [61.6 to 89.4] | 74.1 [61.0 to 89.8]
    Symptoms Score | 87.5 [75.0 to 100.0] | 91.7 [70.8 to 100.0] | 91.7 [70.8 to 100.0]
    Daily Activities Score | 66.7 [45.8 to 89.6] | 65.6 [49.0 to 92.7] | 66.7 [47.9 to 91.7]
    Treatment Concerns Score | 83.3 [66.7 to 94.4] | 80.6 [63.9 to 94.4] | 80.6 [66.7 to 94.4]
    Satisfaction with how well your current treatment controls your AF | 83.3 [66.7 to 100.0] | 83.3 [66.7 to 100.0] | 83.3 [66.7 to 100.0]
    Satisfaction with the extent that treatment has relieved your symptoms of AF | 83.3 [66.7 to 100.0] | 83.3 [66.7 to 100.0] | 83.3 [66.7 to 100.0]
Patient-Reported Outcomes Measurement Information System 29 item instrument (PROMIS-29)-29 [Median (Inter-Quartile Range); unit: Score on a scale] — PROMIS-29 assesses 7 domains (physical function; depression and sadness; pain interference; satisfaction with participation in social roles and activities; fatigue; anxiety and fear; sleep disturbance), 4 questions each. Scores are transformed using a T-score for a mean of 50, standard deviation of 10 in a referent population. Higher scores indicate worse health for the depression, pain, fatigue, anxiety/sleep domains, and better health for the physical function and satisfaction domains. Pain Intensity item is scored 0 (No pain) to 10 (Worst imaginable pain) in the past 7 days.
  Score on a scale
    Physical Function (T-score) | 40.5 [35.6 to 48.3] | 43.5 [36.7 to 57.0] | 41.9 [36.7 to 48.3]
    Anxiety (T-score) | 40.3 [40.3 to 51.2] | 48.0 [40.3 to 56.8] | 48.0 [40.3 to 55.8]
    Depression (T-score) | 41.0 [41.0 to 51.8] | 41.0 [41.0 to 51.8] | 41.0 [41.0 to 51.8]
    Fatigue (T-score) | 51.0 [46.0 to 58.8] | 51.0 [43.1 to 58.8] | 51.0 [46.0 to 58.8]
    Sleep Disturbance (T-score) | 50.5 [43.8 to 56.1] | 50.5 [43.8 to 57.0] | 50.5 [43.8 to 56.1]
    Ability to Participate in Social Roles and Activities (T-score) | 51.9 [44.2 to 64.2] | 51.9 [44.2 to 64.2] | 51.9 [44.2 to 64.2]
    Pain Interference (T-score) | 55.6 [41.6 to 62.5] | 53.9 [41.6 to 61.2] | 53.9 [41.6 to 61.2]
    Pain Intensity (Global07) | 3 [1 to 5] | 3 [1 to 6] | 3 [1 to 6]
Health literacy [Count of Participants; unit: Participants] — The Newest Vital Sign was used to assess health literacy. Scores range from 0 to 6, with limited limited health literacy defined by a score of 0 to 1; possibility of limited literacy by a score of 2 or 3; and adequate health literacy by a sore of 4, 5, or 6.
  Participants
    High likelihood of limited health literacy | 20 | 20 | 40
    Possibility of limited health literacy | 30 | 30 | 60
    Adequate health literacy | 73 | 70 | 143
Brief Health Literacy Screening Instrument [Count of Participants; unit: Participants] — A 4-item, well-validated instrument for health literacy screening with each item scored from 1-5, with higher scores indicating adequate health literacy. Scores from 4-12 suggest limited health literacy; 13-16 moderate health literacy; 17-20 adequate health literacy.
  Participants
    Limited | 7 | 8 | 15
    Moderate | 14 | 27 | 41
    Adequate | 102 | 85 | 187
Patient Health Questionnaire-8 [Median (Inter-Quartile Range); unit: units on a scale] — The Patient Health Questionnaire-8 is an 8-item instrument for depression screening. Scores range from 0 to 24 with higher scores indicating greater likelihood of depression. Scores 5-9 indicate likelihood of mild depression; 10-14, moderate depression; 15-19, moderately severe depression; and 20-24, severe depression.
  units on a scale | 3 [1 to 6] | 3 [1 to 8] | 3 [1 to 7]
Underwent prior electrophysiologic procedure [Count of Participants; unit: Participants] — History of prior electrophysiologic procedures.
  Participants
    Underwent electrical cardioversion: No | 91 | 81 | 172
    Underwent electrical cardioversion: Yes | 32 | 39 | 71
    Underwent medication cardioversion: No | 121 | 118 | 239
    Underwent medication cardioversion: Yes | 2 | 2 | 4
    Underwent a pacemaker insertion: No | 107 | 100 | 207
    Underwent a pacemaker insertion: Yes | 16 | 20 | 36
    Underwent a defibrillator insertion: No | 115 | 110 | 225
    Underwent a defibrillator insertion: Yes | 8 | 10 | 18
    Underwent a pulmonary vein isolation: No | 123 | 120 | 243
    Underwent a pulmonary vein isolation: Yes | 0 | 0 | 0
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: Weight (kg) / Height^2(m^2)] — Body Mass Index (BMI) recorded directly from the electronic health record.
  Weight (kg) / Height^2(m^2) | 31.7 [27.1 to 38.1] | 29.9 [26.3 to 35.6] | 31.2 [26.7 to 37.1]
General Health [Count of Participants; unit: Participants] — Self-reported general health assessment, range 1-5, with higher scores indicating perception of better general health.
  Participants
    Excellent | 5 | 4 | 9
    Very Good | 28 | 32 | 60
    Good | 48 | 47 | 95
    Fair | 34 | 29 | 63
    Poor | 8 | 8 | 16
Smoking History [Count of Participants; unit: Participants]
  Ever smoked cigarettes: No | 49 | 58 | 107
  Ever smoked cigarettes: Yes | 73 | 62 | 135
  Ever smoked cigarettes: Prefer not to respond | 1 | 0 | 1
  Currently smoke: No | 114 | 107 | 221
  Currently smoke: Yes | 8 | 13 | 21
  Currently smoke: Prefer not to respond | 1 | 0 | 1
Montreal Cognitive Assessment [Count of Participants; unit: Participants] — Scores for 76 participants in the intervention arm and 75 participants in the usual care arm were not assessed at baseline, survey was added part way through study recruitment.
  The score for 1 participant in the intervention arm was not assessed due to participant refusing to answer one section of the survey, therefore unable to score the survey.
  Participants
    Score less than 19 | 13 | 8 | 21
    Score greater than or equal to 19 | 33 | 37 | 70
    Not assessed | 77 | 75 | 152

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Days Covered
Description: Proportion of Days Covered (PDC), obtained from collection of electronic prescription and pharmacy fill data, and defined as the proportion of availability of medication for the period of interest, here the period from the date of the baseline to the 12-month examination. PDC range is 0 to 1.00 with higher values indicating greater proportion of days with medication over the 12-month period of study participation as indicated by pharmacy records.
Time Frame: 12 months
Population: Pharmacy data were not available for 8 intervention and 7 usual care participants.
Measure: Median (Inter-Quartile Range); unit: Proportion of days covered
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 115 | 113
Proportion of days covered | 1.0 [0.9 to 1.0] | 0.9 [0.8 to 1.0]
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Proportion of days covered assessed as a continuous measure (range 0-1) at 12 months between study arms adjusted for trial stratification factors (type of anticoagulant treatment). We determined that a sample size of 120 in the intervention group and 120 in the control group enables us to detect a minimum difference in PDC as small as 12.6% with 90% power. Power calculations assume use of 2-sided tests with 0.05 significance level; Test type: Superiority; p = 0.22, t-test, 2 sided — A priori threshold for statistical significance p<0.05

2. Secondary Outcome: Self-reported Non-adherence
Description: Self-reported non-adherence to oral anticoagulation with a 3-item instrument with each item scored 1-5 and lower scores indicating adherence. Scores dichotomized to classify participants as adherent (indicated by reporting 1 on all 3 items) or as non-adherent (indicated by reporting ≥ 2 on any of the 3 items).
Time Frame: 4, 8 and 12 months
Population: Intervention 4-month: n=111 (11 withdrawals [w/d]; 1 missed visit) 8-month: n=109 (total 13 w/d; 1 missed visit) 12-month: n= 108 (total 13 w/d; 2 missed the visit)
  Usual care 4-months: n=107 (10 w/d; 3 missed visit) 8 months: n=107 (total 10 w/d; 3 missed visit) 12-months: n=103 (total 12 w/d; 5 missed visit)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 123 | 120
Participants
  4 Month: number analyzed (Participants) | 111 | 107
  4 Month: Adherent | 99 | 87
  4 Month: Non-adherent | 12 | 20
  8 Month: number analyzed (Participants) | 109 | 107
  8 Month: Adherent | 99 | 87
  8 Month: Non-adherent | 10 | 20
  12 Month: number analyzed (Participants) | 108 | 103
  12 Month: Adherent | 94 | 85
  12 Month: Non-adherent | 14 | 18

3. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS)-29
Description: Measure Description: Patient-Reported Outcomes Measurement Information System (PROMIS)-29 assesses 7 domains (physical function; depression and sadness; pain interference; satisfaction with participation in social roles and activities; fatigue; anxiety and fear; sleep disturbance), 4 questions each, and Pain Intensity with a single item. The 7 domain scores are transformed using a T-score with a mean of 50, standard deviation of 10, in a referent population. Higher scores indicate worse health for the depression, pain, fatigue, anxiety/sleep domains, while higher scores indicate better health for the physical function and satisfaction domains. The single Pain Intensity item is scored 0 (No pain) to 10 (Worst imaginable pain) in the past 7 days.
  Further details on PROMIS scoring are available at https://www.healthmeasures.net/images/PROMIS/manuals/PROMIS_Adult_Profile_Scoring_Manual.pdf.
Time Frame: 4, 8, and 12 months
Population: Intervention arm:
  4-month: n=111 (11 withdrawals [w/d]; 1 missed visit) 8-month: n=109 (total 13 w/d; 1 missed visit) 12-month: n=108 (total 13 w/d; 2 missed visit)
  Usual Care:
  4-month: n=107 (10 w/d; 3 missed visit) 8-month: n=107 (total 10 w/d; 3 missed visit) 12-month: n=103 (total 12 w/d; 5 missed visit)
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 123 | 120
Score on a scale
  Physical Function: 4 month: number analyzed (Participants) | 111 | 107
  Physical Function: 4 month | 41.9 [35.6 to 48.3] | 41.9 [36.7 to 57.0]
  Physical Function: 8 month: number analyzed (Participants) | 109 | 107
  Physical Function: 8 month | 41.9 [36.7 to 48.3] | 41.9 [35.6 to 57.0]
  Physical Function: 12 month: number analyzed (Participants) | 108 | 103
  Physical Function: 12 month | 41.9 [36.7 to 48.3] | 43.5 [36.7 to 57.0]
  Anxiety: 4 month: number analyzed (Participants) | 111 | 107
  Anxiety: 4 month | 40.3 [40.3 to 53.7] | 48.0 [40.3 to 55.8]
  Anxiety: 8 month: number analyzed (Participants) | 109 | 107
  Anxiety: 8 month | 40.3 [40.3 to 53.7] | 48.0 [40.3 to 55.8]
  Anxiety: 12 month: number analyzed (Participants) | 108 | 103
  Anxiety: 12 month | 40.3 [40.3 to 53.7] | 40.3 [40.3 to 53.7]
  Depression: 4 month: number analyzed (Participants) | 111 | 107
  Depression: 4 month | 41.0 [41.0 to 51.8] | 41.0 [14.0 to 51.8]
  Depression:8 month: number analyzed (Participants) | 109 | 107
  Depression:8 month | 41.0 [41.0 to 49.0] | 41.0 [41.0 to 51.8]
  Depression: 12 month: number analyzed (Participants) | 108 | 103
  Depression: 12 month | 41.0 [41.0 to 51.8] | 41.0 [41.0 to 51.8]
  Fatigue: 4 month: number analyzed (Participants) | 111 | 107
  Fatigue: 4 month | 51.0 [46.0 to 57.0] | 53.1 [43.1 to 58.8]
  Fatigue: 8 month: number analyzed (Participants) | 109 | 107
  Fatigue: 8 month | 51.0 [46.0 to 57.0] | 51.0 [43.1 to 58.8]
  Fatigue: 12 month: number analyzed (Participants) | 108 | 103
  Fatigue: 12 month | 48.6 [46.0 to 57.0] | 48.6 [43.1 to 57.0]
  Sleep Disturbance: 4 month: number analyzed (Participants) | 111 | 107
  Sleep Disturbance: 4 month | 48.4 [43.8 to 54.3] | 50.5 [41.1 to 56.1]
  Sleep Disturbance: 8 month: number analyzed (Participants) | 109 | 107
  Sleep Disturbance: 8 month | 48.4 [41.1 to 54.3] | 50.5 [43.8 to 56.1]
  Sleep Disturbance: 12 month: number analyzed (Participants) | 108 | 103
  Sleep Disturbance: 12 month | 48.4 [43.8 to 54.3] | 50.5 [41.1 to 56.1]
  Ability to Participate in Social Roles and Activities: 4 month: number analyzed (Participants) | 111 | 107
  Ability to Participate in Social Roles and Activities: 4 month | 51.9 [44.2 to 64.2] | 51.9 [44.2 to 64.2]
  Ability to Participate in Social Roles and Activities: 8 month: number analyzed (Participants) | 109 | 107
  Ability to Participate in Social Roles and Activities: 8 month | 51.9 [44.2 to 58.3] | 51.9 [44.2 to 58.3]
  Ability to Participate in Social Roles and Activities: 12 month: number analyzed (Participants) | 108 | 103
  Ability to Participate in Social Roles and Activities: 12 month | 51.0 [44.2 to 58.3] | 51.9 [44.2 to 64.2]
  Pain Interference: 4 month: number analyzed (Participants) | 111 | 107
  Pain Interference: 4 month | 57.1 [41.6 to 62.5] | 55.6 [41.6 to 61.2]
  Pain Interference: 8 month: number analyzed (Participants) | 109 | 107
  Pain Interference: 8 month | 55.6 [41.6 to 61.2] | 55.6 [41.6 to 61.2]
  Pain Interference: 12 month: number analyzed (Participants) | 108 | 103
  Pain Interference: 12 month | 55.6 [41.6 to 61.2] | 55.6 [41.6 to 62.5]
  Pain Intensity (Global 07): 4 month: number analyzed (Participants) | 111 | 107
  Pain Intensity (Global 07): 4 month | 4 [1 to 63] | 3 [1 to 6]
  Pain Intensity (Global 07): 8 month: number analyzed (Participants) | 109 | 107
  Pain Intensity (Global 07): 8 month | 3 [1 to 5] | 3 [1 to 5]
  Pain Intensity (Global 07): 12 month: number analyzed (Participants) | 108 | 103
  Pain Intensity (Global 07): 12 month | 4 [2 to 6] | 3 [1 to 6]

4. Secondary Outcome: Atrial Fibrillation Effect on Quality of Life (AFEQT)
Description: The Atrial Fibrillation Effect on Quality of life (AFEQT) is a widely used measure of atrial fibrillation-specific health-related quality of life. Scores range from 0 to 100 with higher scores indicating superior health-related quality of life in AF.
Time Frame: 4, 8 and 12 months
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 123 | 120
score on a scale
  4 Month: number analyzed (Participants) | 111 | 107
  4 Month | 77.8 [61.1 to 93.5] | 79.6 [60.2 to 92.6]
  8 Month: number analyzed (Participants) | 109 | 107
  8 Month | 79.6 [65.7 to 91.7] | 77.8 [63.9 to 91.7]
  12 Month: number analyzed (Participants) | 108 | 103
  12 Month | 76.9 [66.2 to 92.6] | 82.4 [62.0 to 92.6]

5. Secondary Outcome: Emergency Room (ER) Visits and Hospitalizations
Description: The number of emergency room visits and hospitalizations quantified at 12 months.
Time Frame: 12 months
Population: Intervention:
  n=112 (11 withdrawals prior to month-4 visit, date of first collection of this outcome)
  Usual care n=110 (10 withdrawals prior to month-4 visit, date of first collection of this outcome)
Measure: Number; unit: ER visits or hospitalization events
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 112 | 110
ER visits or hospitalization events | 71 | 163

6. Secondary Outcome: Days of Hospitalization
Description: The number of days of hospitalization ascertained from extraction of electronic health records through the 12 months of study duration. Total days spent in hospital over 12 months were summarized as a single count for each participant.
Time Frame: 12 months
Population: as for outcome 5
Measure: Number; unit: days
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 112 | 110
days | 292 | 638

ADVERSE EVENTS:
Time Frame: Data collection occurred from date of consent through the participants 12-month visit.
Description: The study team learned of Adverse Events and Serious Adverse Events by participant interviews at the 4-, 8-, and 12-month assessments; direct contact by participants during scheduled check-in calls; review of the electronic health record; communication from referring physicians or participants' providers; or contact with study team initiated by family or other participant surrogates.
Arm/Group | Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 2/123 | 2/120
Serious Adverse Events (participants affected / at risk) | 30/123 | 26/120
Other Adverse Events (participants affected / at risk) | 18/123 | 26/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=123) | Usual Care (N=120)
Heart failure (Cardiac disorders) | 16 (18) | 12 (21)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 7 (12)
Chest pain-cardiac (Cardiac disorders) | 4 (4) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (2)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
COVID-19 (General disorders) | 3 (3) | 3 (3)
Death NOS (General disorders) | 2 (2) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Ambulatory dysfunction (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute upper GI bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 2 (2)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 2 (2)
Movements involuntary (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Intracranial hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hematruia (Renal and urinary disorders) | 0 (0) | 1 (1)
Suprapubic catheter dislodged (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
Medication side effect (Investigations) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Non-small cell lung cancer resection (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=123) | Usual Care (N=120)
Chest pain-cardiac (Cardiac disorders) | 0 (0) | 2 (6)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 3 (3)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Elevated blood pressure (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 2 (5)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bleeding varicose vein (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Impaired mobility (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 1 (1) | 0 (0)
Right leg pain (General disorders) | 0 (0) | 1 (1)
Shortness of breath (General disorders) | 0 (0) | 1 (1)
Viral syndrome (General disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (3)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1)
Joint infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Floaters (Eye disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT04075994/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT04075994/ICF_001.pdf